CLINICAL TRIAL: NCT02233413
Title: Low Level Light Therapy (LLLT) With Near Infrared Light Emitting Diodes in Patients With Moderate Traumatic Brain Injury (TBI)
Brief Title: Light Therapy for Moderate Traumatic Brain Injury
Acronym: LLLT for TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rajiv Gupta, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2013P000430; W81XWH-13-2-0067 CDMRP (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-06-05; First posted 2014-09-08 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Moderate Traumatic Brain Injury (TBI)
Keywords: Traumatic brain injury; TBI; Low-level light therapy; LLLT; LLLT helmet
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-active LLLT helmet application (Sham Comparator): A helmet containing near infrared LED's (LLLT helmet) will be applied to the head, however, the LEDs will not be turned on / activated.
  Interventions: Device: Non-active LLLT helmet application
- Active LLLT helmet application (Active Comparator): A helmet containing near infrared LEDs (LLLT helmet) will be applied and the LEDs will be turned on/activated
  Interventions: Device: Active LLLT helmet application

INTERVENTIONS:
Device: Active LLLT helmet application — LED helmet applied with light activated
  Arms: Active LLLT helmet application
Device: Non-active LLLT helmet application — LED helmet applied without light activated
  Arms: Non-active LLLT helmet application

SUMMARY:
The purpose of this research study is to find out if a specialized helmet that provides low levels of near infrared light, also known as low-level light therapy (LLLT) has any effect on the recovery of people who have recently (within 72h) suffered a moderate traumatic brain injury (TBI).

DETAILED DESCRIPTION:
The specific aim of this pilot study is to determine the feasibility of using the LLLT helmet in patients with moderate TBI and to quantify the response to LLLT using magnetic resonance (MR) and clinical outcome measures. We hypothesize that we will be able to quantify the response to LLLT through MR imaging and clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Injury within 72 hours at the time of consent;
* Head injury requiring hospital admission;
* A Glasgow Coma Scale (GCS) score of 9-12 or 13-15 with abnormal imaging.

Exclusion Criteria:

* Need for emergency neurosurgical intervention (including placement of intracranial pressure monitoring devices or drainage catheters);
* Hemodynamic instability as determined by the clinician;
* History of any of the following: (i) brain tumor; (ii) prior TBI occurring within the past year and requiring hospital admission; (iii) a new diagnosis within the past year of either stroke or epilepsy; (iv) an established diagnosis of any of the following neurodegenerative diseases: Alzheimer's, Picks, Parkinson's, Lewy body dementia, Huntington's, amytropic lateral sclerosis, spinocerebellar ataxia, vascular dementia, HIZ-associated dementia, dementia due to metabolic causes (Addison, Cushing, hypothyroidism, renal failure, prophyrias, Wilson, mitochondrial diseases, Wernicke-Korsakoff syndrome, and dementia of unknown etiology.
* Pregnancy (all women of child-bearing age will need to have a negative pregnancy test prior to the start of the interventional portion of the study);
* Electrical implants such as cardiac pacemakers or perfusion pumps;
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants, or any other contra-indications to MRI.
* Clinical determination that subject cannot undergo MRI
* Breastfeeding
* Unstable cervical fractures
* Scalp lacerations or surgical wounds severe enough to preclude safe application of device
* Unreliable to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-06; Primary Completion 2019-07-31 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Gupta, MD, PhD, Principal Investigator — Massachusetts General Hospital; Benjamin Vakoc, PhD, Study Director — Massachussetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chan ST, Mercaldo N, Figueiro Longo MG, Welt J, Avesta A, Lee J, Lev MH, Ratai EM, Wenke MR, Parry BA, Drake L, Anderson RR, Rauch T, Diaz-Arrastia R, Kwong KK, Hamblin M, Vakoc BJ, Gupta R. Effects of Low-Level Light Therapy on Resting-State Connectivity Following Moderate Traumatic Brain Injury: Secondary Analyses of a Double-blinded Placebo-controlled Study. Radiology. 2024 May;311(2):e230999. doi: 10.1148/radiol.230999. PMID 38805733
- [Derived] Figueiro Longo MG, Tan CO, Chan ST, Welt J, Avesta A, Ratai E, Mercaldo ND, Yendiki A, Namati J, Chico-Calero I, Parry BA, Drake L, Anderson R, Rauch T, Diaz-Arrastia R, Lev M, Lee J, Hamblin M, Vakoc B, Gupta R. Effect of Transcranial Low-Level Light Therapy vs Sham Therapy Among Patients With Moderate Traumatic Brain Injury: A Randomized Clinical Trial. JAMA Netw Open. 2020 Sep 1;3(9):e2017337. doi: 10.1001/jamanetworkopen.2020.17337. PMID 32926117

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-active LLLT Helmet Application | Active LLLT Helmet Application
Started | 35 | 33
Completed | 24 | 19
Not Completed | 11 | 14
Not completed — Lost to Follow-up | 7 | 9
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-active LLLT Helmet Application | Active LLLT Helmet Application | Total
Number analyzed (Participants) | 24 | 19 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.00 (14.68) | 46.05 (19.93) | 50.49 (17.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Injury Mechanism [Count of Participants; unit: Participants]
  Bike/Motorcycle Accident with Helmet | 4 | 0 | 4
  Bike/Motorcycle Accident without Helmet | 0 | 1 | 1
  Fall | 14 | 11 | 25
  Other | 1 | 0 | 1
  Pedestrian accident with car/motorcycle/bike | 3 | 1 | 4
  Restrained Automobile Accident | 0 | 3 | 3
  Unrestrained Automobile Accident | 1 | 0 | 1
  Violence/assault | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety and Feasibility of Applying Light Therapy After Moderate TBI
Description: Number of subjects to successfully complete light therapy without serious unanticipated adverse events related to application of the device.
Time Frame: up to seven days after enrollment
Population: Subjects who completed light or sham treatment and at least one MRI scan. 43 patients completed the study with at least one MRI scan, 19 subjects in the Light treatment group and 24 subjects in the sham treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-active LLLT Helmet Application | Active LLLT Helmet Application
Number analyzed (Participants) | 24 | 19
Participants | 24 | 19

2. Secondary Outcome: Neuroreactivity of Light Therapy to the Injured Brain Based on MRI Using the Fazekas Scale for Periventricular White Matter (PVWM)
Description: The presence of chronic white matter disease was evaluated using Fazekas scale. The scale divides the white matter in periventricular and deep white matter, and each region is given a grade depending on the size and confluence of lesions.
  periventricular white matter (PVWM). 0 = absent
  1. = "caps" or pencil-thin lining
  2. = smooth "halo"
  3. = irregular periventricular signal extending into the deep white matter
  A neuroradiologist evaluated the 3D T2-SPACE-FLAIR images to detect the presence of T2 hyperintensities and their degree (0: absent; 1: mild; 2: moderate; and 3: severe) for PVWM. Higher values represent a worse outcome.
Time Frame: up to 3 months after treatment
Population: Of the 68 patients that were randomized, 28 completed at least one light therapy session. 43 patients completed the study with at least one MRI scan. 19 subjects in the light treatment group and 24 subjects in the sham treatment group. One MRI was deemed low quality and excluded from analysis (19 light treatment / 23 sham)
Measure: Count of Participants; unit: Participants
Arm/Group | Non-active LLLT Helmet Application | Active LLLT Helmet Application
Number analyzed (Participants) | 23 | 19
Participants
  PVWM: Absent / "Caps" or pencil-thin lining (1) | 19 | 18
  PVWM: Smooth "halo" (2) | 3 | 1
  PVWM: Irregular periventricular signal (3) | 1 | 0

3. Secondary Outcome: Neuroreactivity of Light Therapy to the Injured Brain Based on MRI Using the Fazekas Scale for Deep White Matter (DWM)
Description: The presence of chronic white matter disease was evaluated using Fazekas scale. The scale divides the white matter in periventricular and deep white matter, and each region is given a grade depending on the size and confluence of lesions.
  deep white matter (DWM) 0 = absent
  1. = punctate foci
  2. = beginning confluence
  3. = large confluent areas
  A neuroradiologist evaluated the 3D T2-SPACE-FLAIR images to detect the presence of T2 hyperintensities and their degree (0: absent; 1: mild; 2: moderate; and 3: severe) for DWM. Higher values represent a worse outcome.
Time Frame: up to 3 months after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Non-active LLLT Helmet Application | Active LLLT Helmet Application
Number analyzed (Participants) | 23 | 19
Participants
  DWM: Absent(0)/Puctuate foci(1) | 19 | 16
  DWM: Beginning confluence (2) | 3 | 3
  DWM: Large confluent areas | 1 | 0

4. Secondary Outcome: Neuroreactivity of Light Therapy to the Injured Brain Based on Neurcognitive Function
Description: RPQ is a 16 item self-assessment questionnaire completed via an in-person or phone interview. Each item in the questionnaire is assessed on a 5-point scale ranging from 0 (no problem) - 4 (severe problem). The questions are grouped in two non-overlapping sets: the RPQ-3 includes early, objective, physical symptoms, and the RPQ-13 group includes later, more cognitive and behavioral symptoms. The RPQ-3 encompasses headache, dizziness, and nausea/vomiting. The RPQ-13 includes questions evaluating noise sensitivity, sleep disturbance, fatigue, irritability, depressed mood, forgetfulness, poor concentration, longer thinking time, blurred vision, light sensitivity, double vision, and restlessness. The RPQ-3 ranges from 0 - 12 (best to worst) and RPQ-13 ranges from 0 - 52 (best to worst). RPQ Total is the theoretical max/min RPQ score with a combined possible score ranging from 0-64 (best to worst). The outcome measures are
Time Frame: RPQ scores were collected at approx 72 hours, 14 days, 3 months, and 6 months and the mean was calculated for the values reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-active LLLT Helmet Application | Active LLLT Helmet Application
Number analyzed (Participants) | 24 | 18
score on a scale
  RPQ-3 | 4.55 (3.13) | 3.94 (3.19)
  RPQ-13 | 12.64 (7.83) | 10.94 (9.98)
  RPQ-Total | 17.18 (10.01) | 14.88 (12.08)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed during study enrollment through study completion, an average of 1 year.
Arm/Group | Non-active LLLT Helmet Application | Active LLLT Helmet Application
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 7/31 | 4/28
Other Adverse Events (participants affected / at risk) | 20/31 | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-active LLLT Helmet Application (N=31) | Active LLLT Helmet Application (N=28)
Operation for tibial & fibular fracture (Surgical and medical procedures) | 0 (0) | 1 (1) — Severe, unexpected, unrelated. Subject came back for scheduled operation due to nonunion left distal tibial & fibular fracture
Subdural hematoma (Nervous system disorders) | 1 (1) | 0 (0) — Severe, expected, unrelated. During data review a SDH was discovered on study MRI which was not present on clinical CT.
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) — Severe, unexpected, unrelated. Subject came back to hospital due to pancreatitis
MSSA bacteremia (Infections and infestations) | 1 (1) | 0 (0) — Severe, unexpected, unrelated. Subject went back to hospital due to MSSA bacteremia
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Severe, unexpected, unrelated. Subject went back to hospital due to COPD exacerbation.
Hospital visit due to headache (Nervous system disorders) | 3 (3) | 0 (0) — Severe, expected, unrelated.
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Severe, unexpected, unrelated. Subject went back to hospital due to suicidal ideation in the setting of intermittent depressive symptoms over years, chronic pain, and other difficulties. Evaluated and cleared by psychiatry.
Hemorrhagic cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) — Severe, unexpected, unrelated. Subject went back to hospital due to hemorrhagic cystitis.
Rectal foreign body (Surgical and medical procedures) | 1 (1) | 0 (0) — Severe, unexpected, unrelated. Subject went back to hospital due to rectal foreign body
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-active LLLT Helmet Application (N=31) | Active LLLT Helmet Application (N=28)
Symptom reporting (Nervous system disorders) | 13 (13) | 10 (10) — Reporting of one or more of the following: Headache, blurred vision, double vision, dizziness, numbness, NV, ringing, noise, light, forgetfulness, thinking, concentrating, irritable, frustrated, restless, sleeping, fatigue, depressed.
Persistent cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Subject visited urgent care for persistent cough
Numbness/tingling in toes (Nervous system disorders) | 0 (0) | 1 (1) — Subject reported numbness/tingling in toes 1 week to 3 month time point
Glass from motor vehicle accident removed (Surgical and medical procedures) | 1 (1) | 0 (0) — Subject went back to hospital to have glass from motor vehicle accident removed from skin on forehead.
Broken nose (Surgical and medical procedures) | 1 (1) | 0 (0) — Subject went back to hospital to have broken nose corrected.
Fracture repair (Surgical and medical procedures) | 1 (1) | 0 (0) — Subject went back to hospital for repair of zygomaticomaxillary complex (ZMC) and orbital floor fractures.
Alcohol abuse (Social circumstances) | 0 (0) | 1 (6) — Subject went back to hospital due to alcohol abuse/intoxication.
Musculoskeletal neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject went back to hospital due to neck pain.
Fall (Social circumstances) | 1 (1) | 0 (0) — Subject went back to hospital due to fall
Dislocated shoulder (Surgical and medical procedures) | 0 (0) | 1 (1) — Subject went back to hospital for dislocated shoulder
Cataract surgery (Eye disorders) | 0 (0) | 1 (2) — Subject went back to hospital for cataract surgery
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Subject went back to hospital due to dizziness
Shoulder sprain (Surgical and medical procedures) | 1 (1) | 1 (1) — Subject returned to hospital due to motor vehicle accident with diagnosis of shoulder sprain
Hemorrhagic cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Hemorrhagic cyst

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT02233413/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT02233413/SAP_001.pdf